CLINICAL TRIAL: NCT01774058
Title: The Intraoperative Arterial Measurement of the Blood Flow Volume After Iloprost Stimulation in Diabetics and Non-diabetics: Implication for Outcome-prediction and Perioperative Therapy
Brief Title: The Arterial Measurement of the Blood Flow Volume After Iloprost Stimulation
Acronym: ILOFLOW
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prim PD Dr Afshin Assadian (Other)
Collaborators: Wilhelminenspital Vienna (Other)
Responsible Party: Sponsor-Investigator, Prim PD Dr Afshin Assadian, Prim PD Dr, Wilhelminenspital Vienna
Organization: Wilhelminenspital Vienna (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILOFLOW2.0
Record Dates: First submitted 2013-01-07; First posted 2013-01-23 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Diabetes; Arteriosclerosis; Peripheral Arterial Occlusive Disease; Neuropathy
Keywords: blood flow volume; ilomedin; measurement; intraarterial; neuropathy
MeSH Terms: conditions — Diabetes Mellitus; Arteriosclerosis; Peripheral Arterial Occlusive Disease 1 | interventions — Solvents; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ilomedin, bloodflow volume, measurement, (Experimental): Surgery was performed under general anesthesia via a longitudinal skin incision. After systemic administration of 5000 IU of unfractionated Heparin, the peripheral vessels were clamped. Following a longitudinal arteriotomy, thrombendarterectomy of the common femoral artery was performed in all cases, extending into the deep femoral artery and superficial femoral artery when necessary. At the end of the reconstruction, 3000 ng of iloprost (Ilomedin), diluted in 15ml saline solution, were administered into the common femoral artery. Distal to the injection site doppler flow measurement was performed at the common femoral artery prior to arteriotomy, prior to the intraarterial application of iloprost and 5 and 10 minutes afterwards, using the Sono TT FlowLab instrument. During the procedure, systemic arterial blood pressure was continuously documented using a pressure transducer connected to an intraarterial cannula placed in the radial artery of the forearm.
  Interventions: Drug: Ilomedin

INTERVENTIONS:
Drug: Ilomedin — 3000ng ilomedin in 15ml salt water will be injected intraarterial into the common femoral artery over 2 minutes for one time,then the investigators will measure the blood flow volume after 5 and then after 10 minutes on the common femoral artery. The patients will be observed by the anaesthesiologist. The patient will get ilomedin one day before the surgery and then for 6 day after surgery into the vein. (10microgramm/o,5ml in 250ml salt water)
  Other Names: Product Code 1-22460; ATC Code: B01AC11; concentrate and solvent for injection

SUMMARY:
A prospective case-control study was performed to investigate the effect of iloprost on the intraoperative flow volume in diabetic and non-diabetic patients as well as the effect of peripheral neuropathy in patients with peripheral arterial occlusive disease (PAOD) undergoing arterial reconstruction (primary endpoint).

100 patients undergoing femoral artery reconstruction or femorodistal bypass surgery were included. Prior to surgery, peripheral nerve conduction velocity was measured. Blood flow volume at the common femoral artery was assessed using a Doppler flowmeter (Sono TT FlowLab; ) before reconstruction, prior to the intraarterial application of 3000ng of iloprost and 5 and 10 minutes afterwards. Peripheral resistance units (PRU) were calculated as a function of mean systemic arterial pressure (MAP) and flow volume (VF): PRU = MAP (mmHg) / VF (ml/min).

DETAILED DESCRIPTION:
The therapeutic properties of prostanoids appear to be primarily due to its vasodilative effect. However, the inhibition of platelet aggregation with a limitation of thrombus formation and the inhibition of the adhesion of leucocytes to endothelial lesions also help to improve blood flow in the peripheral circulation .

It is currently unclear which effects of prostanoids are predominant for diabetic patients. The present study was performed to assess potential differences of iloprost efficiency for patients with or without type II diabetes mellitus with or without peripheral neuropathy.

The study was a single center, controlled, non- randomized interventional study. All patients provided their written consent. The study has been approved by the Ethics Committee of the city of Vienna in 2012 (EC nr: 11-144-0512) and was extended annually for the last two years. Performance of the study complied with the World Medical Association Declaration of Helsinki regarding ethical conduct of research involving human subjects.

The study was designed to enroll 100 consecutive patients with peripheral arterial occlusive disease undergoing surgical reconstruction of the inguinal arteries and/or femorodistal bypass surgery. Indication for surgery included PAOD Fontaine stage IIb (waking distance less than 200 meters), III (rest pain) or IV (tissue loss). Surgical procedures were planned and the absence of inflow stenoses verified based on MRI or CT angiography. Exclusion criteria for participation in the study comprised contraindications for the application of iloprost as well as a planned spinal anesthesia. Patients were divided into two groups based on being diabetic type II or non-diabetic. Before surgery measurement of nerve conduction velocity was performed by a trained nurse at the Department of Physiotherapy in order to determine the presence of neuropathy.

Surgery was performed under general anesthesia via a longitudinal skin incision. After systemic administration of 5000 IU of unfractionated Heparin, the peripheral vessels were clamped. After longitudinal arteriotomy, thrombendarterectomy of the common femoral artery was performed in all cases, extending into the deep femoral artery and superficial femoral artery when necessary. In some cases, this was followed by femoropopliteal bypass surgery. Provided the systolic blood pressure was equal to or above 100 mmHg at the end of the reconstruction, 3000 ng of iloprost (Ilomedin), diluted in 15ml saline solution, were injected into the common femoral artery. Distal to the injection site doppler flow measurement was performed at the common femoral artery prior to arteriotomy, prior to the intraarterial application of iloprost, 5 and 10 minutes afterwards, using the Sono TT FlowLab instrument (em-Tec GmbH, Munich). Transmission heads were selected to fit tightly around the reconstructed vessel without producing a stenosis. During the procedure, systemic arterial blood pressure was continuously documented using a pressure transducer connected to an intraarterial cannula placed in the radial artery of the forearm. The result of the arterial reconstruction was routinely checked by intraoperative on- table angiography. Before discharge from the hospital the surgical reconstruction was controlled by duplex ultrasound as well as an assessment of the ankle brachial index.

Statistical analysis was performed with SPSS 15.0 for Windows (SPSS Inc, Chicago, Ill). To correct all measurements of flow volume for blood pressure, peripheral resistance units (PRU) were calculated as a function of mean systemic arterial pressure (MAP) and flow volume (VF): PRU = MAP (mmHg) / VF (ml/min).

The patient population was stratified by the presence of diabetes and by the presence of peripheral neuropathy in the operated limb. Kolmogorov-Smirnov testing confirmed normal distribution of all continuous variables. Descriptive statistics (mean, standard deviation, range) were applied to acquired data, and tests for dependent or independent variables were used for comparison of continuous variables, as applicable. Categorical variables were expressed as frequencies and percentages, and differences between groups were investigated by the Pearson Chi -square and Fisher exact tests. Patient characteristics potentially modulating the effect of iloprost were investigated by linear regression analysis. P values < 0.05 were considered significant.

ELIGIBILITY:
Inclusion Criteria:

* patients with diabetes and non diabetes
* patients with peripheral artery occlusive disease and who undergo surgical treatment in distal vessels
* spinal anesthesia
* written consent

Exclusion Criteria:

* pregnancy
* heart attack the last 6 months
* stroke the last 6 months
* hypotension
* edema of the lungs
* heart failure
* heart disease
* chronic obstructive pulmonary disease (COPD)
* ulcus ventriculi
* renal disease
* coronary disease
* immaturity
* general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-10; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
The measurement of the blood flow volume is done with the Sono TT FlowLab (em-Tec GmbH, Munich) ultrasound instrument on the common femoral artery in diabetics and non-diabetics after ilomedin administration. | 6 weeks after surgery
  Before surgery reconstruction the first measurement with the Sono TT FlowLab (em-Tec GmbH, Munich) ultrasound instrument will be done on the common femoral artery and then after surgery reconstruction. Therefore there will be different measuring heads exactly fitting around the vessels. Then the administration of 3000ng Ilomedin® in 15ml saline will be injected into the common femoral artery via a a cannula over two minutes if the systolic blood pressure of the patient is over 100mm Hg. The blood flow volume will be measured again after five and ten minutes on the same point. Those results will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Assadian, Prim PD Dr, Principal Investigator — Georg Hagmüller Institute for Vascular Research Wilhelminenhospital Vienna, Austria
Locations (1):
- Department of vascular and endovascular surgery, Georg Hagmüller Institute for Vascular Research Wilhelminenhospital, Vienna, Austria